CLINICAL TRIAL: NCT04877717
Title: An Open-Label, Single-Arm, Multi-Center Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of SHR-A1904 in Patients With Advanced Solid Tumors
Brief Title: A Study of SHR-A1904 in Patients With Advanced Solid Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1904-I-101
Record Dates: First submitted 2021-04-27; First posted 2021-05-07 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Cancer

STUDY DESIGN:
Intervention Model Description: SHR-A1904 monotherapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A1904 (Experimental)
  Interventions: Drug: SHR-A1904

INTERVENTIONS:
Drug: SHR-A1904 — SHR-A1904

SUMMARY:
The study is being conducted to assess the safety and tolerability of SHR-A1904 in patients with advanced solid cancer and to determine the dose-limiting toxicity (DLT), maximum tolerated dose (MTD), and recommended phase II dose (RP2D) of SHR-A1904

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study
2. Males or females aged 18-75 years old
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
4. Has a life expectancy≥ 3 months
5. Has at least one measurable lesion as defined by RECIST v1.1
6. Pathologically confirmed advanced solid cancer

Exclusion Criteria:

1. Plan to receive any other anti-tumor treatments during the study treatment period of this study
2. Received other clinical investigational products or treatments within 4 weeks before the first dose of the study
3. Received anti-tumor therapies such as chemotherapy, radiotherapy, biological therapy, targeted therapy, or immunotherapy within 4 weeks before the first dose of the study
4. Underwent a major surgery other than diagnosis or biopsy within 4 weeks before the first dose of the study
5. Subjects with known brain metastases
6. Grade II-IV cardiac insufficiency as per the New York Heart Association (NYHA) criteria; arrhythmia requiring long-term drug control; unstable angina or acute myocardial infarction within 6 months before the first dose of the study
7. presence of accompanying diseases (such as poorly controlled hypertension, serious diabetes mellitus, thyroid disorder, psychosis, etc.) that may pose serious risks to the safety of the subject or may affect the subject's ability to complete the study, or any other situation as judged by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Determine the Maximum Tolerated Dose of SHR-A1904 | up to 1 year

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | up to 1 year
Time to maximum concentration (Tmax) | up to 1 year
Area under the drug concentration-time curve from time 0 to the last measurable concentration time point (AUC0-t) | up to 1 year
Anti-drug antibody (ADA) of SHR-A1904 | up to 1 year
Objective response rate (ORR) | up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Ruan DY, Wu HX, Luo SX, Huang WW, Liang XJ, Niu ZX, Dang Q, Li HL, Pan ZY, Lu HX, Zhang YQ, Li XY, Xiao XY, Cai SR, Dong YG, Zhang J, Li Z, Lan HT, Wang X, Zhou Y, Liu L, Liu HL, Xu PS, Suo AL, Jia RN, Li YQ, Peng XD, Wang SC, Yu AA, Xie J, Qiu MZ, Xu RH. The antibody-drug conjugate SHR-A1904 for targeting CLDN18.2 in advanced gastric or gastroesophageal junction cancer: a phase 1 trial. Nat Med. 2025 Sep;31(9):3037-3046. doi: 10.1038/s41591-025-03781-w. Epub 2025 Jul 16. PMID 40670772